CLINICAL TRIAL: NCT06126120
Title: Prevalence, Determinants, and Challenges of Adherence With Colonoscopy Check-up in People With Lynch Syndrome: a Questionnaire-based Study
Brief Title: Colonoscopy Check-up in People With Lynch Syndrome
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 329468
Record Dates: First submitted 2023-11-03; First posted 2023-11-13 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Lynch Syndrome
Keywords: Lynch Syndrome; Colonoscopy; Surveillance
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lynch Syndrome, an inherited condition, increases bowel cancer risk. People with Lynch Syndrome are recommended to have regular colonoscopies where a camera in a tube is used to look inside the bowel for cancer and for polyps (growths that sometimes can become cancerous). UK guidelines recommend that people with Lynch Syndrome have colonoscopy check-up every 2 years after reaching a certain age; however, they face many challenges which make it difficult to have the recommended check-up.

Among a subset of people with Lynch Syndrome in England, this study will investigate the:

* percentage who are having colonoscopy check-up as recommended by UK guidelines
* factors influencing whether a person is more/less likely to have the recommended colonoscopy check-up
* views, experiences, and challenges of living with Lynch Syndrome and colonoscopy check-up

This study will collect information from people in the 'Lynch Syndrome registry pilot' using a questionnaire. The Cancer Screening and Prevention Research Group (CSPRG) at Imperial College London are conducting the Lynch Syndrome registry pilot, which is recruiting people with Lynch Syndrome who are aged >18 years and in the Cancer Prevention Programme 3 (CaPP3) trial, from Nov 2022-Nov 2023.

This study will include people in the Lynch Syndrome registry pilot who provided consent on the registry pilot consent form to be contacted about future research and are aged ≥25 years. People who have had previous surgery to remove their rectum will be excluded.

The investigators will use the 'Views, experiences, and challenges of colonoscopy check-up' questionnaire, together with a few pieces of additional information previously collected as part of the Lynch Syndrome registry pilot.

Participation involves completing the questionnaire only. The study will take approximately one year from administering the questionnaire to sharing results with participants.

ELIGIBILITY:
Inclusion Criteria:

* People in the Lynch Syndrome registry pilot who have provided consent to be contacted about future research and are aged ≥25 years

Exclusion Criteria:

* People who have had surgery involving removal of their rectum

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include people who are in the Lynch Syndrome registry pilot and meet the eligibility criteria for the present study. The Lynch Syndrome registry pilot is recruiting people with Lynch Syndrome who are aged >18 years and in the CaPP3 trial.
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Participant non-adherence to 2-yearly colonoscopy check-up. | 1 day
  Participant non-adherence to 2-yearly colonoscopy check-up will be assessed on a single occasion, considering participants' three most recent colonoscopy check-ups, measured as a percentage.

SECONDARY OUTCOMES:
The four most important challenges to having colonoscopy check-up for participants. | 1 day
  The four most important challenges to having colonoscopy check-up will be assessed on a single occasion, considering participants' responses in the questionnaire. The questionnaire asks participants to select their most important challenges from a given list, and the top four selections will be considered the most important challenges.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda J Cross, PhD, Principal Investigator — Imperial College London
Locations (1):
- Cancer Screening and Prevention Research Group (CSPRG), Department of Surgery and Cancer, Queen Elizabeth The Queen Mother (QEQM) Building, St Mary's Hospital, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No